CLINICAL TRIAL: NCT01024049
Title: Identification Of Blood Markers For Asymptomatic Ventricular Dysfunction
Acronym: IBLOMAVED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C06-15
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Heart Failure
Keywords: heart failure blood left ventricular dysfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — plasma sample blood RNA sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Asymptomatic LVD: patients over 18 years old with patients with cardiovascular risk (obesity, diabetes, dyslipidemia, arterial hypertension, age, gender, familial history) and asymptomatic left ventricular dysfunction (LVD).
- healthy controls: individuals over 18 years old free of disease and treatments.
- patients with cardiovascular risk: patients with cardiovascular risk (obesity, diabetes, dyslipidemia, arterial hypertension, age, gender, familial history)
- chronic heart failure patients: patient with chronic heart failure
- acute heart failure patients: acute heart failure patients

SUMMARY:
The diagnosis of asymptomatic left ventricular dysfunction is difficult in general practice since it requires transthoracic cardiac echocardiography that is generally performed in specialized services. Although blood BNP levels monitoring can be of some help in heart failure diagnosis is is mostly a late biomarker that is secreted upon heart stretch and has many limitations. Therefore the aim of this study is to identify new specific blood biomarkers that would help for asymptomatic left ventricular dysfunction diagnosis in large populations with cardiovascular risk.

DETAILED DESCRIPTION:
Recognition of asymptomatic left ventricular dysfunction (ALVD) and early stages of heart failure (HF) are a diagnostic challenge for physicians. Patient history and physical examination may fail to provide a definitive diagnosis; additional testing are required to aid in diagnosis. More than 20 million people worldwide are estimated to have HF. Despite recent therapeutic advances, morbidity and mortality after the onset of heart failure remain high (35 % at 5 years after diagnosis). In addition, the annual cost of heart failure is estimated to be greater than that of myocardial infarction and all cancers combined. Consequently, prevention of heart failure through identification and management of risk factors and preclinical phases of the disease is a priority. Clearly identification of asymptomatic patients is difficult but would prevent further development of HF by initiation of early adapted medical and non medical treatment.

We propose to search for markers of ALVD, in patients that have cardiovascular risk factors. These new biomarkers should be earlier, more specific and more accurate than the one that we already have such as B-type natriuretic peptide (BNP), which is the most recently, established. BNP has been clearly associated with HF but is a relatively late stage marker for HF and is not specific for HF. In addition BNP has been shown to be a poor marker in obese or diabetic patients. Therefore the need of early specific biomarkers for LVD before HF is irreversibly initiated is strong.

We propose to compare blood samples from 5 groups of patients carefully defined: 1) without cardiovascular risk factors ; 2) With cardiovascular risk factors and without ALVD; 3) With cardiovascular risk factors and with ALVD. 4) chronic heart failure patients ; 5) Acute heart failure patients. Groups will be matched for risk factors and treatments.

Three distinct approaches will be performed: - A transcriptomics one that will monitor white blood cell transcriptome ; a proteomic one that will use high throughput SELDI-TOF profiling and a metabolic profiling one using Nuclear Magnetic Resonance.

ELIGIBILITY:
Inclusion Criteria (5 groups defined):

Patients with Obesity or diabetes or arterial hypertension with or without : acute or chronic heart failure, left ventricular hypertrophy, left ventricular dysfunction symptomatic or not.

Healthy control patients

Exclusion Criteria:

cancer and/or other other severe chronical or infectious pathologies. Patient is unable to sign or understand the consent form Patients is on any dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy individuals
  2. Patients with cardiovascular risk
  3. Patients with cardiovascular risk and asymptomatic left ventricular dysfunction
  4. Chronic heart failure patients
  5. Acute heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Galinier, MD-PHD, Principal Investigator — Hospital of Toulouse, INSERM
Locations (1):
- Hospital from Toulouse Rangueil, Pr Galinier department (Cardiology A), Toulouse, Midi-Pyrénées, France

REFERENCES:
- [Derived] Rouet K, Rouet P, Koukoui F, Galinier M. Diagnostic accuracy and rapid testing of a novel acute heart failure biomarker: A laboratory evaluation and comparison with natriuretic peptides. Ann Clin Biochem. 2025 Aug 28:45632251378035. doi: 10.1177/00045632251378035. Online ahead of print. PMID 40877033
- [Derived] Koukoui F, Desmoulin F, Galinier M, Barutaut M, Caubere C, Evaristi MF, Murat G, De Boer R, Berry M, Smih F, Rouet P. The prognostic value of plasma galectin-3 in chronic heart failure patients is maintained when treated with mineralocorticoid receptor antagonists. PLoS One. 2015 Mar 18;10(3):e0119160. doi: 10.1371/journal.pone.0119160. eCollection 2015. PMID 25786035